CLINICAL TRIAL: NCT06263569
Title: Effectiveness of Total Hip Arthroplasty for Patients With Osteoarthritis, a Target Trial Emulation Study
Acronym: EAGLE
Status: Completed | Type: Observational
Sponsor: JointResearch (Other)
Responsible Party: Principal Investigator, Rudolf Poolman, Prof. dr., JointResearch
Other Study IDs: SDB 2023-002
Record Dates: First submitted 2024-01-12; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Total hip arthroplasty (THA): Total hip arthroplasty surgery
  Interventions: Procedure: Total hip arthroplasty
- Non-Total hip arthroplasty (THA): No total hip arthroplasty surgery performed / control group.

INTERVENTIONS:
Procedure: Total hip arthroplasty — Unilateral primary total hip arthroplasty procedure.
  Groups: Total hip arthroplasty (THA)

SUMMARY:
The aim of this study is to assess the effect of total hip arthroplasty on hip disability and pain compared to non-surgery in patients with hip osteoarthritis, using target trial emulation to emulate a randomized controlled trial.

DETAILED DESCRIPTION:
The ideal research design to investigate effectiveness of total hip arthroplasty (THA) would be to randomize patients between surgery and (delayed) non-surgery. Such a randomized controlled trial (RCT) is deemed unethical due to the effect size of THA shown in observational studies.

In this study a target trial is specified (a randomized controlled trial between THA and non-THA) and the target trial is emulated using observational data of 2 dutch hospitals participating in the value based health care (VBHC) programme for hip osteoarthritis. The objective of this study is to compare the effect of THA surgery on hip disability and pain between patients that did or did not receive THA surgery during the Covid-19 pandemic. It is hypothesized that THA is effective in restoring hip function and reduction of pain compared to the control group. The effect of THA has not been demonstrated by means of an RCT before. This study can contribute to the available evidence by assessing causal effectiveness of THA by means of RCT target trial emulation.

As a secondary aim, the assumption of pseudo-random group allocation will be assessed. Logistic regression analysis will be used to test whether group allocation is independent of patient characteristics (age, sex, HOOS-PS baseline, NRS baseline, physical therapy before baseline and follow-up time.

ELIGIBILITY:
Inclusion Criteria:

* Patients on the waiting list for primary THA between 1-4-2020 up until 31-3-2022 in OLVG or Martini hospital.
* Completed intake questionnaire (HOOS-PS baseline)
* Indication osteoarthritis of the hip

Exclusion Criteria:

* Patients that received THA on both sides within follow-up (1-4-2020 and 1-1-2022) will be excluded.
* Patients with other indications than osteoarthritis of the hip were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hip osteoarthritis, eligible for primary total hip arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Hip disability and Osteoarthritis Outcome Score Physical function Short form (HOOS-PS), change score from baseline | 3 months
  Ranging from 0 (no difficulty) to 100 (extreme difficulty)

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) pain during weight bearing, change score from baseline | 3 months
  Ranging from 0 (no pain) to 10 (worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Poolman, Prof., Principal Investigator — OLVG
Locations (1):
- OLVG, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT06263569/Prot_SAP_000.pdf